CLINICAL TRIAL: NCT04221022
Title: PHYSICAL ACTIVITY AS COPING STRATEGY FOR ACADEMIC STRESS AMONG UNDERGRADUATE FEMALE COLLEGIATE STUDENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zohra Institute of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZIHS-1272/MS/05
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Physical Activity and Stress
Keywords: Physical Activity; academic stress; Light Physical activity; Moderate Physical Activity; Vigorous Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Light physical activity (Group 1) (Active Comparator): Female collegiate students were assessed by using Academic stress scale questionnaire, Cohen Perceived stress Scale and rapid assessment of physical activity (RAPA) to determine physical activity level and academic stress. They were assigned into Light Physical activity. Each subject in first group completed 6 weeks of exercise sessions which aimed to cope up academic stress among female collegiate students. Each subject was evaluated for changes in symptoms in each week.
  Interventions: Other: Light physical activity
- Moderate physical activity (Group 2) (Active Comparator): Female collegiate students were assessed by using Academic stress scale questionnaire, Cohen Perceived stress Scale and rapid assessment of physical activity (RAPA) to determine physical activity level and academic stress. They were assigned into moderate Physical activity. Each subject in first group completed 6 weeks of exercise sessions which aimed to cope up academic stress among female collegiate students. Each subject was evaluated for changes in symptoms in each week.
  Interventions: Other: Moderate physical activity
- Vigorous physical activity (Group 3) (Active Comparator): Female collegiate students were assessed by using Academic stress scale questionnaire, Cohen Perceived stress Scale and rapid assessment of physical activity (RAPA) to determine physical activity level and academic stress. They were assigned into vigorous Physical activity. Each subject in first group completed 6 weeks of exercise sessions which aimed to cope up academic stress among female collegiate students. Each subject was evaluated for changes in symptoms in each week.
  Interventions: Other: Vigorous physical activity

INTERVENTIONS:
Other: Light physical activity — Each session started with leisure walk, duration of which was set to 35 minutes. Frequency set for the session was that each individual of the group had to walk for five days a week for total of six weeks. (total 30 days in six weeks)
  Arms: Light physical activity (Group 1)
Other: Moderate physical activity — Each session started with brisk walk, duration of which was set to 30 minutes. Frequency set for the session was that each individual of the group had to walk for five days a week for total of six weeks. (total 30 days in six weeks)
  Arms: Moderate physical activity (Group 2)
Other: Vigorous physical activity — Each session started with jogging, duration of which was set to 15 minutes. Frequency set for the session was that each individual of the group had to walk for five days a week for total of six weeks. (total 30 days in six weeks)
  Arms: Vigorous physical activity (Group 3)

SUMMARY:
Physical Inactivity is one of the major cause causing academic stress in students, so effectiveness of Light, moderate and vigorous physical activity as a baseline treatment were assessed through academic stress scale questionnaire, Cohen Perceived stress Scale and rapid assessment of physical activity (RAPA).

DETAILED DESCRIPTION:
A total of 388 students participated in first phase of study and total 60 students with moderate academic stress were filtered. Among those only 37 were physically inactive from last one month by the assessment through RAPA (Rapid assessment of physical activity). ASS (Academic stress scale), Cohen Perceived stress Scale and RAPA questionnaires were used to collect data. Three equally distributed groups were given three different modes of physical activities i.e light, moderate & vigorous.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate female students between 18-24 years.
* Students with moderate level of academic stress
* Students inactive from last one month

Exclusion Criteria:

* Students with any other type of stress
* Students with other psychological disorders
* Student with known systemic disease.
* Physically active from last one month were excluded.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All female participants
Enrollment: 37 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Academic stress scale | upto 6 weeks
  it helps in measuring the level of academic stress experienced by college students due to five types of sources viz. Personal Inadequacy, Interactions with Peers and Teachers, Fear of Examination, Inadequate Facilities at College and Parents Expectations and SES.
Rapid Assessment Physical Activity scale | upto 6 weeks
  Physical activity level of the patients was also observed through rapid assessment of physical activity with categories as "0" for No involvement and "1" for yes and the results showed that those who are involved in any type of physical activity have a better functional outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Syed Alamdar Hussain, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR